CLINICAL TRIAL: NCT00215852
Title: A Randomized, Dose-Ranging Study of Alferon® LDO [Low Dose Interferon Alfa-n3 (Human Leukocyte Derived)] in Asymptomatic HIV+ Subjects
Brief Title: A Randomized, Dose-ranging Study of Alferon LDO in Asymptomatic HIV+ Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: AIM ImmunoTech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LDO-101
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-08

CONDITIONS: HIV Infections
Keywords: Alferon LDO; Low Dose Oral Interferon; Alfa-n3; Human Leukocyte Derived; HIV; Asymptomatic HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): 500 IU
  Interventions: Drug: Alferon LDO
- 2 (Active Comparator): 1000 IU
  Interventions: Drug: Alferon LDO
- 3 (Active Comparator): 2000 IU
  Interventions: Drug: Alferon LDO

INTERVENTIONS:
Drug: Alferon LDO — 500 IU, taken orally each evening, for 10 consecutive days while holding in the mouth for at least 2 minutes prior to swallowing, for 10 daysday 5 of each 28 day cycle.

SUMMARY:
To conduct a randomized dose-ranging study to evaluate the safety and activity of orally administered low dose interferon alfa-n3 as an immunomodulator in subjects with asymptomatic HIV-1 infection. The primary endpoints of the study will include an increase or upregulation in genes known to be mediators of interferon response. Secondary endpoints will include the absolute CD4 count and plasma HIV RNA levels.

DETAILED DESCRIPTION:
This study will be an open-label, randomized outpatient study in HIV infected subjects using a range of doses of Alferon LDO. The first nine (9) patients enrolled will not be randomized. Instead, the first three (3) patients will receive 500 IU, the second three (3) patients will receive 1000 IU, and the final three (3) patients will receive 2000 IU. Once three (3) patients at a given dose level have received at least 8 doses without grade 3 toxicity, patients may be enrolled at the next higher dose level. Following enrollment of the first nine (9) patients, additional patients will be randomized to receive one of the three (3) dose levels of Alferon® LDO. The Alferon LDO (natural interferon alfa-n3) will be in a buffer solution and taken orally once each day for 10 consecutive days at doses equal to 500 IU, 1000 IU, or 2000 IU.

Pretherapy baseline evaluations will be performed within the three (3) week period prior to randomization.

Drug will be dispensed for a ten day treatment period, during which time any clinical symptoms and adverse events will be evaluated. Laboratory samples (2.5 ml blood) for microarray analysis evaluations will be made twice during baseline and 12-14 hours following doses 1, 4, and 10 on study days 2, 5, and 11, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. HIV-1 plasma RNA > 500 copies/ml (Roche Amplicor assay) or similar assay within 45 days of starting oral dosing.
3. Karnofsky performance status of 100
4. Subjects must be asymptomatic with regard to HIV related clinical symptoms including the following opportunistic infections: Oral candidiasis (thrush), cutaneous herpes simplex, fever, diarrhea, weight loss ≥ 10% of body weight, seborrheic dermatitis, chronic mucocutaneous fungal infections or Kaposi's sarcoma. Subjects with a history of AIDS are not eligible.
5. Serum creatinine ≤ 1.5 ULN; serum bilirubin ≤ 2.0 ULN.
6. Total WBC ≥ 3000/mm3, platelet count ≥ 100,000/mm3 and granulocytes ≥ 1500 mm3.
7. Absolute CD4 cell count greater than 400 (based on the average CD4 count from the two pretherapy tests).
8. Hemoglobin > 10.0 g/dl.
9. AST < 4 times upper normal limit.
10. ALT < 4 times upper normal limit.
11. Serum Albumin > 2.0 g/dl.
12. Written informed consent.
13. Females must either be of non-child bearing potential, or utilize an effective form of contraception and have a negative pregnancy test within 14 days of entry.
14. For those subjects who are on antiretroviral therapy, they must have been on a stable dose schedule for at least 90 days prior to study entry and must continue on the same schedule during the treatment phase of this study.

Exclusion Criteria:

1. Pregnant or nursing women, or women not using an effective form of contraception.
2. Less than 18 years of age.
3. Active IV drug users.
4. Absolute CD4 ≤ 400 mm3 (based on the average CD4 counts from the two pretherapy tests).
5. Receipt of any immunosuppressive agent, chemotherapy, or systemic steroids within 45 days of study entry.
6. Receipt of any immunomodulator such as BCG vaccine, isoprinosine, or similar experimental agents within 45 days of study entry.
7. Evidence of chronic hepatitis, or other active gastrointestinal, renal, respiratory, endocrine, hematologic, cardiovascular, neurological, or psychiatric disorder that would limit the subject's ability to complete the study period.
8. Unlikely or unable to comply with the requirements of the protocol.
9. Patients unwilling or unable to give informed consent.
10. Patients on any other concurrent experimental medication.
11. Concurrent, chronic prophylactic use of any systemic antifungal medication (e.g. ketoconazole, fluconazole, clotrimazole) or of any systemic anti-viral (e.g. acyclovir or ganciclovir) except for antiretroviral therapy.
12. Patients using any form of interferon therapy during the 6 weeks prior to study entry. If prior interferon therapy has been received, the subject must not have known development of antibodies to interferon.
13. Hospitalized subjects, or those with an active viral infection other than HIV, within 2 weeks of study entry.
14. Transfusion dependent subjects (subjects requiring > 1 unit of packed RBC per month within the 3 months prior to study entry).
15. Subjects who are symptomatic of their HIV infection at study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Gene expression analysis | Days 0, 2, 5, 11, 12 and 16

SECONDARY OUTCOMES:
CD4 Level | Days 0, 11 and 16

CONTACTS AND LOCATIONS:
Overall Officials: David R Strayer, MD, Study Director — AIM ImmunoTech Inc.
Locations (2):
- United States (2):
  - Drexel University School of Medicine, Philadelphia, Pennsylvania
  - Philadelphia FIGHTS, Philadelphia, Pennsylvania